CLINICAL TRIAL: NCT01008072
Title: Ultra-rapid Opiate Detoxification Using Deep Sedation and Prior Oral Buprenorphine Preparation.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Murat Bahar, Assaf-Harofeh MC
Other Study IDs: 173/09
Record Dates: First submitted 2009-11-04; First posted 2009-11-05 (Estimated); Last update posted 2009-11-05 (Estimated); Status verified 2009-11

CONDITIONS: Opioid Addiction
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- without buprenorphine preparation
- with buprenorphine preparation

SUMMARY:
The methods of detoxification under general anesthesia have been criticized because of limited data on safety and long-term follow-up. Premedication with buprenorphine has been advocated to improve safety. In current study we want to evaluate the importance of buprenorphine preparation in rapid opioid detoxification process, under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Opioid addiction

Exclusion Criteria:

* Age < 18 Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All opioid addicted patients who wants to undergo rapid detoxification under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-12; Primary Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesiology department, Assaf-Harofeh MC, Beer-Yaakov, Zrifin, Israel